CLINICAL TRIAL: NCT00580086
Title: Monitoring Response to Neoadjuvant Chemotherapy by the Use of Breast Proton MR Spectroscopy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Laura Liberman, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 06-146
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; MR spectroscopy; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1
  Interventions: Other: MR spectroscopy

INTERVENTIONS:
Other: MR spectroscopy — (1H MRS) on 1.5 Tesla (1.5T), using a software package from General Electric Medical Systems, Milwaukee, WI

SUMMARY:
This study is being done to evaluate if MR spectroscopy will give us more information about whether or not your chemotherapy will work for you. Spectroscopy is a special set of pictures taken with Magnetic Resonance Imaging (MRI) that gives us information about the chemical composition of your breast cancer.

DETAILED DESCRIPTION:
The study aim is to perform MR Spectroscopy (1H MRS) on 1.5 Tesla (1.5T), using a software package from General Electric Medical Systems, Milwaukee, WI on 115 patients with biopsy proven adenocarcinoma of the breast, who will be receiving neoadjuvant chemotherapy as per standard therapeutic protocol, prior to surgical management. The spectroscopic data will be analyzed to determine whether this can enable early prediction of therapeutic response as assessed by RECIST and ultimately surgical pathology after the completion of the full course of drug treatment. The 1H MRS, which is performed at baseline, prior to treatment, halfway through and at the end of the chemotherapy course, just prior to surgery, will be added to the routine MRI examination for the affected breast. Since chemotherapy courses vary in length, the exact timeline will depend on the specific course given. 1H MRS will add 10 minutes to the routine MRI examination, but will not involve additional injections of contrast. In addition, we will perform two extra MRIs combined with 1H MRS examinations for the affected breast, one set the day after and the second set one week after the initiation of chemotherapy. The MRI and 1H MRS will be performed at Memorial Sloan-Kettering Cancer Center, 1275 York Avenue, NY, NY 10021 or at any offsite of MSKCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be ≥ 18 years of age
* Patients with biopsy confirmed adenocarcinoma of the breast, scheduled to receive neoadjuvant chemotherapy prior to surgical management.

Exclusion Criteria:

* Patients who would normally be excluded from undergoing an MRI examination include:

  * Patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field
  * Patients who are pregnant
* Patients who are unable to comply or complete the MRI exam such as patients with claustrophobia and patients who have electrically, magnetically, or mechanically activated implants, such as heart pacemakers, certain types of artificial joints, inner ear implants, eye implants, or certain surgical clips used in vascular surgery.
* Patients who are not candidates for neoadjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are asked to take part in this study because they have breast cancer and are scheduled to receive chemotherapy treatment before having surgery.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The spectroscopic data will be analyzed to determine whether this can enable early prediction of therapeutic response as assessed by RECIST and ultimately surgical pathology after the completion of the full course of drug treatment. | The 1st MRI before start chemotherapy, the 2nd MRI half way through treatment, and the final MRI before surgery. Two MRI exams will be for research only.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Liberman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org